CLINICAL TRIAL: NCT00087685
Title: A Phase II Study of RAD001 in Patients With Recurrent Endometrial Cancer
Brief Title: RAD001 in Recurrent Endometrial Cancer Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2004-0002; NCI-2012-01308 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2004-07-12; First posted 2004-07-14 (Estimated); Results first posted 2016-02-05 (Estimated); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Endometrial Cancer
Keywords: Recurrent Endometrial Cancer; Endometrial; Endometrioid; RAD001; Uterine Cancer
MeSH Terms: conditions — Endometrial Neoplasms; Uterine Neoplasms | interventions — Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- RAD001 (Experimental): RAD001 10 mg by mouth Daily
  Interventions: Drug: RAD001

INTERVENTIONS:
Drug: RAD001 — 10 mg by mouth Daily

SUMMARY:
The goal of this clinical research study is to learn if RAD001 can shrink or slow the growth of tumors in patients who have recurrent endometrial cancer. The safety of this drug will also be studied.

Objectives:

Primary Objective:

1. To determine the efficacy of RAD001 in patients with progressive or recurrent endometrial cancer.

Secondary Objective:

1. To determine the nature and degree of toxicity of RAD001 in this cohort of patients.
2. To characterize, in pre- and post- treatment tumor samples, when available, expression levels of total and phosphorylated mTOR (mammalian "target of rapamycin") as well as relevant upstream and downstream signaling components (optional).

DETAILED DESCRIPTION:
RAD001 is a new drug that was designed to block proteins that are important in the development and growth of cancer.

Before treatment starts, you will have a complete physical exam, routine blood tests (about 2-3 teaspoons), a chest x-ray, and a CT scan or MRI of the abdomen and pelvis. Women who are able to have children must have a negative blood pregnancy test.

Routine blood tests (about 2 teaspoons) will be done weekly during treatment, and before each course of therapy, which is every 4 weeks. A complete checkup including evaluation of side effects, will also be done before each course of therapy and at the end of therapy (4 weeks after treatment ends).

You will take RAD001 10 mg by mouth every day. One course of therapy is 4 weeks long. RAD001 should be taken the same time every day on an empty stomach (fasting state) or after no more than a light, fat-free meal. You should wait at least 6 hours after a eating a regular (not fat-free meal) before taking RAD001. You should not eat fatty foods for at least one hour after taking RAD001.

If side effects occur at this dose, your doctor may lower the RAD001 dose, depending on the severity of the side effects. After an additional 4 weeks of therapy, if the dose was reduced and the side effects have resolved, your doctor may increase the dose back to the original dose, or you may continue at the reduced dose.

You will only be given the amount of drug needed for one course of therapy at a time. You will keep a diary during the study that will list when and how much drug you took. This diary will be reviewed after each course of therapy by the research nurse or physician and filed in your chart.

You will have CT or MRI scans and chest x-rays (only in patients with chest disease) to evaluate the response of your tumor to treatment. These scans will be done after the first two courses (eight weeks) and every third course (every 12 weeks) and at the end of therapy. Treatment will be stopped if the disease gets worse or intolerable side effects occur.

This is an investigational study. RAD001 has been authorized by the FDA for use in research only. Up to 35 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed progressive or recurrent endometrial cancer (endometrioid or mixed with endometrioid component histology; any grade).
2. Patients may have failed no more than two prior chemotherapies for the recurrent disease (does not include chemosensitizing radiation).
3. All patients must have measurable disease. Measurable disease is defined as lesions that can be measured by physical examination or by means of imaging techniques. Ascites and pleural effusions are not considered measurable disease.
4. Patients must have a pretreatment granulocyte count (i.e., segmented neutrophils + bands) of >/=1,500/Fl, a hemoglobin level of >/=9.0 gm/dL and a platelet count of >/=100,000/Fl.
5. Patients must have an adequate renal function as documented by serum creatinine </=2.0 mg/dL.
6. Patients must have adequate hepatic function as documented by a serum bilirubin </=1.5 mg/dL, regardless of whether patients have liver involvement secondary to tumor. Aspartate transaminase (SGOT) must be </=3x institutional upper limit of normal unless the liver is involved with tumor, in that case the aspartate transaminase must be </=5x institutional upper limit of normal.
7. Patients must have a Zubrod performance status of 0, 1, or 2.
8. Patients must have signed an approved informed consent.

Exclusion Criteria:

1. Patients who have previously received RAD001 or another mammalian target of rapamycin (mTOR) inhibitor.
2. Patients whose tumors have serous carcinomas, mixed malignant mullerian tumors (MMMT) components or uterine sarcomas.
3. Patients who have isolated recurrences (vaginal, pelvic, or para-aortic) that are amenable to potentially curative treatment with radiation therapy or surgery.
4. Patients with a history of psychiatric disorders that would interfere with consent or follow-up.
5. Patients with a history of myocardial infarction within the previous six months or congestive heart failure requiring therapy.
6. Patients with a history of prior malignancy (except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer) or other cancer for which the patient has been disease-free for at least five years.
7. Pregnant or lactating women. Women of reproductive potential may not participate unless they have agreed to use an effective contraceptive method.
8. Patients with a history of seizures are ineligible. Patients receiving phenytoin, phenobarbital, or other anti-epileptic prophylaxis are ineligible.
9. Patients with any other severe concurrent disease which would make the patient inappropriate for entry into this study, including significant hepatic, renal, or gastrointestinal diseases.
10. Patients with deep venous or arterial thrombosis (including pulmonary embolism) within 6 weeks of study entry.
11. Patients with >/= grade 2 hypercholesterolemia or hypertriglyceridaemia (fasting state), despite lipid lowering therapy should be excluded from entering the study.
12. Patients currently taking any of the medications listed in Appendix A (Patients will be given a listing of these medications at the time of the informed consent).
13. Known hypersensitivity to everolimus, sirolimus or excipients including hydroxytoluene, magnesium stearate, hydroxypropylmethyl-cellulose, crospovidone and lactulose.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2004-06; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen H. Lu, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: June 18, 2004 to March 20, 2008. All recruitment was done at The University of Texas (UT) MD Anderson Cancer Center.
Groups:
- RAD001: 10 mg orally daily/28-day cycles
Period: Overall Study
Arm/Group | RAD001
Started | 35
Completed | 21
Not Completed | 14
Not completed — Adverse Event | 5
Not completed — Non-Compliance | 1
Not completed — Progressive Disease | 5
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Arm/Group | RAD001
Number analyzed (Participants) | 35
Age, Continuous [Median (Full Range); unit: years] | 59 [38 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 35

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Objective Response Plus Stable Disease Rate (CR + PR + SD)
Description: Response determined by tumor assessments from radiological tests or physical examination using Response Evaluation Criteria In Solid Tumors (RECIST). Complete Response (CR): Disappearance of all target and non-target lesions and no evidence of new lesions documented by two disease assessments at least 4 weeks apart. Partial Response (PR): At least 30% decrease in sum of the longest dimensions (LD) of all target measurable lesions taking as reference the baseline sum of LD. Stable Disease (SD): Any condition not meeting the above criteria. The minimum duration for the SD will be 8 weeks. If the participant has stable disease at the time of the first radiographic evaluation, he/she will be considered to have stable disease. Progressive Disease (PD): At least a 20% increase in the sum of LD of target lesions taking as reference the smallest sum LD or the appearance of new lesions within 8 weeks of study entry.
Time Frame: 8 weeks
Population: Of the 35 participants, four (4) were inevaluable due to inadequate treatment on trial.
Measure: Number; unit: participants
Arm/Group | RAD001
Number analyzed (Participants) | 31
participants
  Complete Response (CR) | 0
  Partial Response (PD) | 0
  Stable Disease (SD) | 14
  Progressive Disease (PD) | 17

2. Primary Outcome: Clinical Benefit Rate
Description: Clinical benefit rate (CBR) is defined as the objective response rate plus the proportion of participants with prolonged stable disease (SD), e.g. nonprogression at 20 weeks. Objective response rate (ORR), determined by tumor assessments from radiological tests or physical examination using Response Evaluation Criteria In Solid Tumors (RECIST).
Time Frame: 20 weeks
Population: Of the 35 participants, four (4) were inevaluable due to inadequate treatment on trial.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | RAD001
Number analyzed (Participants) | 31
percentage of participants | 21 [8.3 to 41.0]

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) collected on average every 4 weeks during clinical evaluation from the start of treatment until discontinuation of treatment. Overall AE collection period: July 12, 2004 to August 07, 2008.
Arm/Group | RAD001
Serious Adverse Events (participants affected / at risk) | 25/35
Other Adverse Events (participants affected / at risk) | 35/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RAD001 (N=35)
Death (General disorders) | 12 (12)
Hyperglycemia (Metabolism and nutrition disorders) | 3 (3)
Pain (General disorders) | 3 (3)
Abdominal Pain (Gastrointestinal disorders) | 5 (5)
Nausea (Gastrointestinal disorders) | 6 (6)
Vomiting (Gastrointestinal disorders) | 6 (6)
Dehydration (Gastrointestinal disorders) | 2 (2)
Fever (General disorders) | 5 (5)
Fever Non-Neutropenic (General disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 2 (2)
Hyponatremia (Metabolism and nutrition disorders) | 2 (2)
Fatigue (General disorders) | 2 (2)
Anorexia (Gastrointestinal disorders) | 1 (1)
Asthenia (General disorders) | 2 (2)
Cystitis (Renal and urinary disorders) | 1 (1)
Decreased Platelets (Blood and lymphatic system disorders) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Decreased Hemoglobin (Blood and lymphatic system disorders) | 2 (2)
Confusion (Nervous system disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pneumonitis (Infections and infestations) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1)
Brain Mass (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3)
Dizziness (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Mucositis (Infections and infestations) | 10 (10)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RAD001 (N=35)
Alkaline Phosphatase Elevated (Metabolism and nutrition disorders) | 7
Alopecia (Skin and subcutaneous tissue disorders) | 3
ALT, SGPT (Metabolism and nutrition disorders) | 8
Anorexia (Gastrointestinal disorders) | 19
AST, SGOT (Metabolism and nutrition disorders) | 10
Bilirubin (Metabolism and nutrition disorders) | 1
Blurred Vision (Eye disorders) | 1
Cholesterol, Serum-High (Metabolism and nutrition disorders) | 21
Constipation (Gastrointestinal disorders) | 13
Cough (Respiratory, thoracic and mediastinal disorders) | 5
Creatinine (Metabolism and nutrition disorders) | 2
Dermatology/Skin (Skin and subcutaneous tissue disorders) | 3
Diaphoresis (General disorders) | 1
Diarrhea (Gastrointestinal disorders) | 8
Distension/Bloating (Gastrointestinal disorders) | 1
Dizziness (Nervous system disorders) | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 9
Edema: Head and Neck (Blood and lymphatic system disorders) | 1
Edema: Limb (Blood and lymphatic system disorders) | 1
Elevated LDH (Metabolism and nutrition disorders) | 1
Fatigue (General disorders) | 26
Fever Without Neutropenia (General disorders) | 4
Gastrointestinal (Gastrointestinal disorders) | 1
Hearing (Ear and labyrinth disorders) | 1
Heartburn (Gastrointestinal disorders) | 1
Hemoglobin (Metabolism and nutrition disorders) | 22
Hot Flashes (Endocrine disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 15
Hyperkalemia (Metabolism and nutrition disorders) | 1
Hypermagnesemia (Metabolism and nutrition disorders) | 1
Hypernatremia (Metabolism and nutrition disorders) | 1
Hypertension (Cardiac disorders) | 1
Hypertriglyceridemia (Metabolism and nutrition disorders) | 23
Hyperuricemia (Metabolism and nutrition disorders) | 1
Hypoglycemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 4
Hypomagnesemia (Metabolism and nutrition disorders) | 9
Hyponatremia (Metabolism and nutrition disorders) | 4
INR (Blood and lymphatic system disorders) | 1
Insomnia (Nervous system disorders) | 2
Leukocytes (Blood and lymphatic system disorders) | 19
Lymphopenia (Blood and lymphatic system disorders) | 15
Memory Impairment (Nervous system disorders) | 2
Metabolic/Laboratory (Metabolism and nutrition disorders) | 21
Mood Alteration (Nervous system disorders) | 9
Mucositis, Oral Cavity (Gastrointestinal disorders) | 8 — Clinical
Mucositis, Oral Cavity (Gastrointestinal disorders) | 6 — Symptomatic
Muscle Weakness (Musculoskeletal and connective tissue disorders) | 4
Nail Changes (Skin and subcutaneous tissue disorders) | 1
Nausea (Gastrointestinal disorders) | 24
Neuropathy, Sensory (Nervous system disorders) | 10
Neutrophils (Blood and lymphatic system disorders) | 11
Pain (Abdomen NOS) (Gastrointestinal disorders) | 3
Pain (Back) (Musculoskeletal and connective tissue disorders) | 3
Pain (Bone) (Musculoskeletal and connective tissue disorders) | 1
Pain (Breast) (Musculoskeletal and connective tissue disorders) | 1
Pain (Buttock) (Musculoskeletal and connective tissue disorders) | 1
Pain (Extremity - Limb) (Musculoskeletal and connective tissue disorders) | 2
Pain (Head) (Nervous system disorders) | 10
Pain (Joint) (Musculoskeletal and connective tissue disorders) | 1
Pain (Muscle) (Musculoskeletal and connective tissue disorders) | 1
Pain (NOS) (General disorders) | 4
Pain (Oral Cavity) (General disorders) | 1
Pain (Pelvis) (Musculoskeletal and connective tissue disorders) | 1
Pain (Skin) (Skin and subcutaneous tissue disorders) | 1
Palpitations (Cardiac disorders) | 1
Platelet Increase (Blood and lymphatic system disorders) | 1
Platelet Decrease (Blood and lymphatic system disorders) | 12
Pruritus (Skin and subcutaneous tissue disorders) | 2
Rash/Desquamation (Skin and subcutaneous tissue disorders) | 8
Rhinorrhea (General disorders) | 1
Rigors/Chills (General disorders) | 6
Somnolence (Nervous system disorders) | 1
Sore Throat (General disorders) | 2
Sweating (General disorders) | 3
Taste Alteration (General disorders) | 4
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 1
Vomiting (Gastrointestinal disorders) | 12
Weight Loss (General disorders) | 8
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes